CLINICAL TRIAL: NCT05362071
Title: Cardiometabolic, Functional and Psychosocial Effects of a Remotely Supervised Exercise Program in Individuals With Type 2 Diabetes
Brief Title: Remotely Supervised Exercise Program in Individuals With Type 2 Diabetes
Acronym: RED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55791622.8.0000.5313
Record Dates: First submitted 2022-04-06; First posted 2022-05-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Exercise; Remote exercise; Glicemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blinded, parallel, superiority, controlled trial. Participants males and females with type 2 diabetes mellitus will be allocated to experimental and control groups based on a randomization sequence created in blocks by an independent research assistant with a 1:1 ratio. Allocation concealment will be implemented through a central randomization routine conducted by the same investigator to generate the sequence. The allocation of participants will occur after the completion of baseline outcomes evaluations.
Who Masked: Outcomes Assessor
Masking Description: Masking Description: Blinding will be implemented for the outcome assessors. All tests and questionnaires will be supervised by an evaluator blinded to the participant's group. Due to the type of intervention, the investigator conducting exercise sessions and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote Exercise Group (Experimental): Participants will practice physical exercises twice a week, remotely and under the supervision of an exercise professional, for 12 weeks.
  Interventions: Other: Remote Exercise Group
- Group control (Other): Participants will receive a booklet with recommendations for physical activity from the physical activity guide for the Brazilian population.
  Interventions: Other: Group control

INTERVENTIONS:
Other: Remote Exercise Group — The intervention will have a weekly frequency of two sessions on non-consecutive days during the first six weeks and three sessions on non-consecutive days for the remaining six weeks. The exercise intervention will consist of four 3-week mesocycles. The session's structure will consist of a warm-up, the main part, in which a combined training program will be carried out, consisting of three distinct blocks, and at the end, stretching. Blocks 1 and 2 will consist of three strength exercises with bodyweight and alternative materials and aerobic training. Between blocks 1 and 2, and later in block 3, participants will take a free walk with displacement in the space they have available in their own home. The session will end with stretching exercises for the main muscle groups. The sessions will last 37 to 57 minutes over 12 weeks, with approximately 5 min of warm-up and stretching, and the main part ranging from 27 min to 47 min throughout the intervention.
  Arms: Remote Exercise Group
Other: Group control — Participants allocated to the GC will receive recommendations for the practice of physical activity based on information from three specific chapters of the Physical Activity Guide for the Brazilian Population (2021). The GC will receive through Whatsapp the information that is available in chapters 1, 4, and 5, which address the following topics: "Understanding Physical Activity," "Physical Activity for Adults," and "Physical Activity for the Elderly." If sending via Whatsapp is not possible, the booklet will be printed and delivered to the participant. At the end of the 12 weeks, the same booklet will be made available to IG participants.
  Arms: Group control

SUMMARY:
The present study, characterized as a randomized clinical trial, aims to verify the effects of a remotely supervised exercise program, compared to a control group, on cardiometabolic, functional, and psychosocial outcomes in individuals with type 2 diabetes (DMT2). Males and females with T2DM from the city of Pelotas/RS who meet the study eligibility criteria will participate in the study. Participants will be randomized into the intervention group (IG) and control group (CG). The IG will perform a 12-week exercise program supervised remotely via video call, while GC will receive recommendations for physical activity. Participants will be evaluated at baseline (week 0) and after intervention (week 13). Initially, data for sample characterization, blood pressure, capillary blood glucose, and functional tests will collect during a home visit. In a second moment, participants will be invited to go to a specific laboratory for collecting glycated hemoglobin (HbA1c). Subsequently, a third date will be scheduled to apply self-administered questionnaires (online via GoogleDocs) related to the quality of life, sleep quality, depressive symptoms, emotional stress related to diabetes, level of physical activity, and eating habits. Additionally, acute glycemic responses will be evaluated before and immediately after an exercise session three times throughout the intervention. Capillary blood glucose will be collected in sessions performed in the initial period of mesocycles 1, 2, and 4. At week 13, reassessment will be realized by the same baseline assessors. Over the 12 weeks, a combined training will be carried out with remote supervision. Participants will perform strength exercises at usual and maximum execution speed and aerobic exercises at a rating of perceived effort between 11 and 15 on Borg's scale. The sessions will have a total duration between 37 and 57 min and a weekly frequency of two weekly sessions in the first six weeks and three weekly sessions in the remaining six weeks. Data will be expressed as mean and standard deviation. Data analysis between pre-and post-intervention moments, as well as between groups, will be performed by Generalized Estimated Equations, with Bonferroni post hoc, considering both per-protocol (including participants who meet 70% of frequency in the intervention) and intention to treat analysis (including all randomized participants), assuming an alpha level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Being under medical treatment using oral hypoglycemic agents
* Female and male patients with type 2 diabetes;
* Not be involved with physical exercises in the last three months;
* Being semi-literate.

Exclusion Criteria:

* Make use of insulin;
* History of cardiovascular disease (except drug-controlled high blood pressure);
* Presence of severe autonomic neuropathy, painful peripheral neuropathy or history of foot injuries, proliferative diabetic retinopathy, severe non-proliferative diabetic retinopathy;
* Muscle or joint impairment that precludes performing physical exercises safely
* Lack of internet access

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | Baseline (week 0) to Post-training (week 13)
  Blood samples will be collected to be later performed a laboratory analysis regarding the HbA1c levels of each of the participants.

SECONDARY OUTCOMES:
Systolic blood pressure | Baseline (week 0) to Post-training (week 13)
  Measurements will be performed using a blood pressure monitor (HEM-7320, OMRON, China). Measurement will be performed on each participant's arm, and then two more measures on the arm with the highest value, always with a 1-minute interval between measurements.
Diastolic blood pressure | Baseline (week 0) to Post-training (week 13)
  Measurements will be performed using a blood pressure monitor (HEM-7320, OMRON, China). Measurement will be performed on each participant's arm, and then two more measures on the arm with the highest value, always with a 1-minute interval between measurements.
Capillary blood glucose | Baseline (week 0) to Post-training (week 13), and pre and immediately after an exercise session performed in the initial period of mesocycles 1, 2 and 4, in the IG participants (each mesocycle consists of 3 weeks).
  Capillary blood glucose will be measured from blood samples (0.6 μL of blood) collected from the participants' fingertips using disposable lancets and reagent strips (Guide Accu-Check, São Paulo). After collection, blood samples will be immediately analyzed by a portable glucometer (Guide Accu-Check, Roche, São Paulo, Brazil).
Lower limb strength | Baseline (week 0) to Post-training (week 13)
  Lower limb strength will be measured by the 30-s chair stand functional test. The test will be performed in a chair standard, in which the participants will start seated with the feet flat the floor and the arms over the chest and will be instructed to stand up, standing completely, and soon after returning to the sitting position, repeating the crossed move as fast as possible. as many times as possible during 30s.The number of times the move is performed will be noted as a result of the test.
Upper limb strength | Baseline (week 0) to Post-training (week 13)
  Upper limb strength will be measured by the Arm Curl test functional. The test will be performed in a chair, in which the participants will start seated with their feet flat on the floor and trunk fully leaning on the chair, holding a dumbbell with the dominant hand, 2 kg for women and 4 kg for men. Flexion of the forearm is requested, followed by extension, this movement is repeated for 30 seconds.The number of correctly performed push-ups are counted.
Agility and dynamic balance | Baseline (week 0) to Post-training (week 13)
  Agility and dynamic balance will be measured using the time up and go (TUG) test. The test will start with the participants seated in a chair with a cone positioned in front of them 3 m away. Participants will be instructed to get up from their chair, walk as fast as possible without running, turn around the cone and return to the starting position. The shortest time of two attempts will be noted as a test result. In addition, the test will also be performed at usual walking speed.
Aerobic capacity | Baseline (week 0) to Post-training (week 13)
  To measure the aerobic capacity of the participants, 2 minute step test will be used. The test measures the maximum number of knee raises that the individual can perform in 2 minutes.At the signal, the participant will begin stationary gait (without running), completing as many knee raises as possible within two minutes. The minimum knee height will be at a midpoint between the patella and the anterior superior iliac spine. The evaluator will count the number of elevations of the right knee.
Flexibility | Baseline (week 0) to Post-training (week 13)
  To measure the flexibility of the lower limbs, the sit and reach (bank wells) test will be performed. Participants must be barefoot, then the will sit the base of the box, with the legs extended and together they will place one of the hands on the other and later will raise the arms vertically. When the evaluator gives the signal, the participant will lean the body forward and reach with the fingertips as much as possible on the graduated ruler, without bending the knees and without using rocking movements (insistence), the evaluator will record the result achieved.
Quality of life (QOL) will be verified using the EUROHIS-QOL 8-item index | Baseline (week 0) to Post-training (week 13)
  Quality of life (QOL) will be verified using the EUROHIS-QOL 8-item index. The questionnaire was validated for the Brazilian population (PIRES et al., 2018). It consists of 8 items (general QoL, general health, energy, activities of daily living, self-esteem, social relationships, finances, and home); each item is answered individually, using a Likert-type scale, from 1 to 5 points. The score ranges from 8 to 40. A higher score indicates better individuals' perception of their QOL.
Sleep quality will be verified using the Pittsburgh Sleep Quality Index Self-report Questionnaire | Baseline (week 0) to Post-training (week 13)
  Sleep quality will be verified using the Pittsburgh Sleep Quality Index Self-report Questionnaire (PSQI). The questionnaire includes 19 questions about the individual's perception and five questions about the roommates' perception related to the participant's sleep (if applicable). These questions are grouped into seven components, with scores ranging from zero to three, where higher scores indicate worse sleep quality (BERTOLAZI et al., 2011).
Depressive symptoms | Baseline (week 0) to Post-training (week 13)
  Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). This instrument was validated for the Brazilian population (SANTOS et al., 2013). It consists of nine questions with four answer options, and its purpose is to verify the presence of depressive symptoms in the last two weeks through a Likert-type scale from 0 to 3 points. The questionnaire also has the tenth question, referring to the interference of symptoms in daily life, and, in total, it is possible to have a score from 0 to 27, which indicates that the lower the score, the smaller the depressive symptoms.
Emotional stress related to diabetes | Baseline (week 0) to Post-training (week 13)
  The Brazilian version of the Problem Areas in Diabetes Scale (B-PAID) (GROSS et al., 2007) will be used to analyze the emotional stress related to diabetes and the impact of diabetes and treatment on the study participants' lives. The questionnaire consists of questions focuses on the quality of life and emotional problems associated with living with diabetes and its treatment. A 5-point Likert scale produces a total score ranging from 0-100, where a high score indicates a high level of emotional distress.
Physical activity levels | Baseline (week 0) to Post-training (week 13)
  Physical activity levels will be measured using the International Physical Activity Questionnaire in its short version (IPAQ-C). It consists of eight self-completion questions in different domains: work, leisure, domestic activities, and physical exercise. Data are expressed in minutes, and the metabolic equivalent is calculated (1 MET: 3.5 ml/kg/min) (PARDINIA et al., 2001).
Eating habits | Baseline (week 0) to Post-training (week 13)
  The Food Frequency Questionnaire (FFQ) will be applied to investigate eating habits, as used in a previous study (GERAGE et al., 2017). The questionnaire consists of a list of 16 foods. According to the Brazilian Food Guide guidelines, these foods will be classified into natural/minimally processed foods and processed or ultra-processed foods. The frequency of consumption reported by the participants will generate scores, where higher scores indicate better eating habits.
Subjective perception of well-being | Post-training (week 13)
  The subjective perception of well-being will be analyzed through a simple question: "in your opinion, how much did participation in the project improve your sense of general well-being?". This question will present structured responses based on the 5-point Likert Scale, ranging from "dissatisfied" to "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas; Rodrigo S Delevatti, PhD, Study Director — Federal University of Santa Catarina
Locations (1):
- Federal University of Pelotas, Pelotas, Brazil, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues SN, Delevatti RS, Carvalho MTX, Bullo V, Bergamin M, Alberton CL. Cardiometabolic, functional, and psychosocial effects of a remotely supervised home-based exercise program in individuals with type 2 diabetes (RED study): study protocol for a randomized clinical trial. Trials. 2023 Oct 19;24(1):679. doi: 10.1186/s13063-023-07704-3. PMID 37858161
- See also: Psychometric properties of the EUROHIS-QOL 8-item index (WHOQOL-8) in a Brazilian sample — https://pubmed.ncbi.nlm.nih.gov/29590264/
- See also: Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index — https://pubmed.ncbi.nlm.nih.gov/21145786/
- See also: Sensitivity and specificity of the Patient Health Questionnaire-9 (PHQ-9) among adults from the general population — https://pubmed.ncbi.nlm.nih.gov/24005919/
- See also: Brazilian version of the Problem Areas in Diabetes Scale (B-PAID): validation and identification of individuals at high risk for emotional distress — https://pubmed.ncbi.nlm.nih.gov/17081645/
- See also: QUESTIONÁRIO INTERNACIONAL DE ATIVIDADE FÍSICA (IPAQ): ESTUDO DE VALIDADE E REPRODUTIBILIDADE NO BRASIL — https://rbafs.org.br/RBAFS/article/view/931
- See also: Effectiveness of a Behavior Change Program on Physical Activity and Eating Habits in Patients With Hypertension: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/28682707/
- See also: Development and validation of a functional fitness test for a community-residing adults — https://www.researchgate.net/publication/279569683_Development_and_validation_of_a_functional_fitness_test_for_a_community-residing_adults
- See also: The timed "Up & Go": a test of basic functional mobility for frail elderly persons — https://pubmed.ncbi.nlm.nih.gov/1991946/